CLINICAL TRIAL: NCT03669575
Title: Modulation of Inflammatory Makers by the Supplementation of n7FA for 3 wk, Randomized Placebo Controlled Crossover Study
Brief Title: Omega 7 Oil and Inflammatory Biomarker Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bastyr University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 16-1575
Record Dates: First submitted 2018-08-10; First posted 2018-09-13 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain | interventions — omega-aminoenantic acid

STUDY DESIGN:
Intervention Model Description: Eligible participants are randomly assigned to one of two crossover arms, i.e verum-placebo or placebo-verum sequence. The verum groups are dosed approximately 900 mg a day omega-7 fatty acid, and placebo group contains other fatty acids except for omega-7. After the baseline assessment, a participant is on the supplement bottle for three weeks before re-assessed, and starts the second bottle without a washout period. The participant is re-assessed at the end of the six weeks before exits the study.
Who Masked: Participant, Investigator
Masking Description: The randomization block of four. Participants, research coordinators, and study clinicians are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- omega 7 - placebo (Experimental): Receiving the active first then switch to the placebo after three weeks
  Interventions: Dietary Supplement: omega 7; Dietary Supplement: Placebo
- placebo - omega 7 (Active Comparator): Receiving the placebo first then switch to the active after three weeks
  Interventions: Dietary Supplement: omega 7; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: omega 7 — Three weeks omega 7 fatty acid nutritional supplement, approximately 900 mg/day
Dietary Supplement: Placebo — Three weeks placebo fatty acids approximately 900 mg/day which does not contain omega 7

SUMMARY:
The purpose of the study is to determine whether the palmitoleic acid supplementation can reduce the serum inflammatory biomarkers and low quality of life scores due to musculoskeletal discomfort. The study design is a 2-arm placebo-controlled double blind crossover trial. The randomized sequence of a single crossover is divided into 1:1 and each supplementation is three weeks with no washout in between.

DETAILED DESCRIPTION:
The purpose of the study is to investigate whether or not the supplementation of a particular omega-7 fatty acid decreases the serum biomarkers of inflammation, i.e. highly sensitive C-reactive protein, TNF-alpha and IL-6 of participants who have been experiencing decreased quality of life (QOL) and having elevated these serum markers. The study is placebo-controlled and conducted in a double blinded manner. Participants will be crossed over on supplements (active and placebo) in a random sequence. The total length of a trial is six weeks in which the participants will be asked to maintain stable diet. The baseline blood draw, physical exam, range of motion, QOL and dietary assessment and taking vitals are performed. After the blood test results and/or QOL assessment confirm the eligibility, three weeks supply of the investigational supplement will be mailed or picked up in person. The supplementation is one gel-capusule a day for three weeks. At the end of three weeks, another blood draw, physical exam, range of motion, and QOL assessment are conducted; then the other investigational supplement will be provided. The assessment of the second supplement will occur after another three-week mark. If no adverse reaction is observed and there is no concerns, the participant will be exited from the study.

The goal of enrollment is 50 participants who are between 18 to 99 years old with decreased quality of life and potentially elevated serum markers of inflammation. Volunteers will be randomized by a block of four so at any given moment, one group does not exceed more than three participants. The study takes place at Kenmore campus.

ELIGIBILITY:
Inclusion Criteria: (any of the below)

* baseline CRP 1.0 mg/L or higher
* > 3 months (chronic) musculoskeletal pain/discomfort, which the participant is able to monitor during the course of trial (6 weeks)

Exclusion Criteria:

* Taking narcotic or opioid pain medication
* Unable to monitor NSAID or OTC pain medication quantity
* Unable to visit Kenmore Washington Clinical Research Center for three times
* Objection from his/her primary care doctor
* Employee or family member of Barlines Organics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
CRP (serum) | 3 weeks
  Quantification of the serum hsCRP level during active supplement
Pain/discomfort (self-assessment from 1 - 10) | 3 weeks
  The self-reported level of the musculoskeletal pain/discomfort during active supplement

SECONDARY OUTCOMES:
Omega 7 (plasma) | 3 weeks
  Quantification of the plasma palmitolenic acid (major omega 7 fatty acid) level during the active supplementation
IL-6 (plasma) | 3 weeks
  Quantification of the plasma IL-6 level during the active supplementation
TNFalpha (plasma) | 3 weeks
  Quantification of the plasma TNFalpha level during the active supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Masa Sasagawa, ND, PhD, Principal Investigator — Bastyr University
Locations (1):
- Bastyr University Clinical Research Center, Kenmore, Washington, United States

IPD SHARING:
Plan to Share IPD: No